CLINICAL TRIAL: NCT05759858
Title: A Single-center Study of the Identification and Prognostic Value of Key Genes in Hepatocellular Carcinoma
Brief Title: Identification and Prognostic Value of Key Genes in Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0856
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2022-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Genomes; Prognosis; Gene targeted therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples were restored at -80℃ for 5 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with hepatocellular carcinoma confirmed by pathology.: Patients with hepatocellular carcinoma confirmed by pathology.
  Interventions: Other: None of intervention

INTERVENTIONS:
Other: None of intervention — None of the interventions was applied.

SUMMARY:
To explore the key genes of human and mouse hepatocellular carcinoma, identify the key genes and prognostic markers, and develop small molecule drugs targeting the key genes to treat hepatocellular carcinoma.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the most common solid malignant tumors and the main cause of cancer-related deaths worldwide. About 750000 new cases of liver cancer are diagnosed every year, half of which are in China. The onset of liver cancer is relatively hidden, and there are generally no symptoms in the early stage. When the patient has obvious clinical symptoms, the disease often belongs to the middle and late stages. The first symptom of liver cancer is liver pain, followed by upper abdominal mass. Some patients also showed some complications of liver cirrhosis, such as black stool, hematemesis, jaundice, liver coma, ascites, etc. A few patients were hospitalized due to symptoms caused by metastatic lesions.

At present, the accuracy of detecting HCC is poor, and the common indicators such as AFP have a certain time lag, which cannot detect patients with liver cancer early. thus, there is an urgent need for a new biomarker for the diagnosis and prognosis of liver cancer. Our research focuses on exploring the key genes of human and mouse hepatocellular carcinoma, identifying the key genes and prognostic markers by means of transcriptome sequencing, and developing small molecule drugs targeting the key genes.

High-throughput sequencing technology was used for sequencing analysis to reflect the expression level of mRNA, small RNA, noncoding RNA, or some other markers. After finding the gene difference between the liver cancer sample and the para-cancer sample, relevant immunohistochemical staining was performed to analyze the overall survival time difference between the patients with high-expression genomes and the patients with low-expression genomes. Follow-up cell and animal experiments were carried out to further verify the effect of target genes on the occurrence and development of liver cancer. In the first month after the operation, the patient was followed up at the outpatient clinic to understand the general situation of the patient after the operation, such as diet and appetite, symptom control, such as fever, abdominal pain, and drainage tube removal. One year and three years after the operation, our center will follow up on the patients and re-hospitalization if necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Hepatocellular carcinoma confirmed by pathology;
2. The patient has no combined organic diseases of heart, lung, and kidney, etc;
3. No history of chemotherapy, radiotherapy, upper abdominal surgery, or combined with other tumors;
4. The patient has successfully completed the operation and has complete clinical information and pathological data.

Exclusion Criteria:

1. Patients who have previous history of other tumors or have undergone upper abdominal surgery;
2. Patients with multiple lesions and distant metastasis;
3. Patients who are complicated with organic diseases of important organs such as heart, lung and kidney and cannot tolerate surgery；
4. Patients who are more than 75 years old or less than 18 years old.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffered hepatocellular carcinoma which was confirmed by pathology. Only surgical treatment is applied to patients.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Key gene differences in hepatocellular carcinoma | Through study completion, an average of 1 year.
  Key gene differences in hepatocellular carcinoma explored by RNA-seq.
Overall survival | Through study completion, up to 5 years.
  The time from the beginning of treatment to death (for any reason).
Disease-free survival | Through study completion, up to 5 years.
  The time from the beginning of treatment to death (for any reason).

SECONDARY OUTCOMES:
The incidence and mortality of postoperative hemorrhage, bile leakage and other complications. | Through study completion, up to 5 years.
  The incidence and mortality of postoperative hemorrhage, bile leakage and other complications.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Yan, Doctor, Study Chair — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China; Yang Tian, Doctor, Study Director — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China; Yuancong Jiang, Doctor, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available from the author on reasonable request.